CLINICAL TRIAL: NCT01335711
Title: A Phase II Open-Label, Randomized, Parallel Group, Safety, Tolerability and Efficacy Study of i.m. Administered CHRONVAC-C in Combination With Electroporation Followed by Standard of Care in Chronic Hepatitis C Virus Genotype 1 Infected and Treatment Naïve Subjects
Brief Title: CHRONVAC-C Study Followed by Standard of Care in Chronic Hepatitis C Virus (HCV) Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ChronTech Pharma AB (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVC-202; 2010-022960-10 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IMP_C/C IL28B (Experimental): C/C IL28B subjects to whom IMP will be administrated prior to SOC
  Interventions: Drug: ChronVac-C + SOC
- SOC_C/C IL28B (Active Comparator): C/C IL28B subjects to whom only SOC will be administrated
  Interventions: Drug: SOC
- IMP_non-C/C IL28B (Experimental): non-C/C IL28B subjects to whom IMP will be administrated prior to SOC
  Interventions: Drug: ChronVac-C + SOC
- SOC_non-C/C IL28B (Active Comparator): non-C/C IL28B subjects to whom only SOC will be administrated
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: ChronVac-C + SOC — IMP: I.m. administration of 500 μg plasmid DNA vaccine CHRONVAC-C (solution for injection) administered i.m. in combination with electroporation using MedPulser® DDS on 2 occasions with 4 weeks in between followed by standard of care (SOC) initiation after 14 - 42 days.
  SOC: Peg-IFN-α-2a (180 μg per week) and Ribavirin (1000 mg/day for subjects with a BW of < 75 kg and 1200 mg/day for subjects with a BW of > 75 kg)
  Arms: IMP_C/C IL28B; IMP_non-C/C IL28B
Drug: SOC — SOC: Peg-IFN-α-2a (180 μg per week) and Ribavirin (1000 mg/day for subjects with a BW of < 75 kg and 1200 mg/day for subjects with a BW of > 75 kg)
  Arms: SOC_C/C IL28B; SOC_non-C/C IL28B

SUMMARY:
To explore the effect on early viral kinetics and viral load, and to determine safety, tolerability and anti-viral response for the plasmid DNA vaccine CHRONVAC-C administered i.m. in combination with electroporation followed by standard of care (SOC) in treatment naïve chronic HCV genotype 1 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 - 65 years of age with a known chronic hepatitis C infection, being treatment naїve (that is not being earlier treated for HCV infection) and a planned start of standard of care within 12 weeks from screening.
* Known genotype 1 infection.
* Viral load equal to 1000 IU/ml or more
* BMI less than 35.
* Considered probable that the deltoid muscles (left and right) of the subject will be reached at vaccination using a 12.7 mm cannula for injection and a 15 mm applicator tip for electroporation.
* Written informed consent obtained, and a copy provided to the subject.
* Subject legally competent and able to communicate effectively with the study personnel.
* Subject likely to co-operate and attend the clinic at the appointed times during the study

Exclusion Criteria:

* Subject having clinically significant concomitant diseases other than HCV in the medical history to the discretion of the investigator.
* Subject having clinically significant findings on physical examination, vital signs, ECG or clinical laboratory evaluations to the discretion of the investigator.
* Subject having clinical or biochemical signs of cirrhosis.
* Positive hepatitis B surface antigen (HBsAg).
* Positive HIV antigen or antibody test.
* Subject having an ongoing and/or known viral infection other than HCV that requires treatment and/or special medical intention.
* Subject having received previous treatment for HCV.
* Radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to the first dose of study drug.
* Treatment with immunomodulating agents such as systemic corticosteroids, IL-2, IFN-alpha, IFN-beta, IFN-gamma within 4 weeks prior to the first dose of study drug. (Corticosteroid nasal sprays, inhaled steroids for asthma and/or topical steroids are allowed, however not on the vaccination area.)
* Immunization within 30 days of the first dose of the study drug.
* Subject having received an investigational drug product, or been enrolled in other investigational drug protocols within a period of 30 days prior to receiving the first dose of the study drug.
* Prior treatment with DNA therapy.
* Known allergy towards vaccines.
* Known allergy or contraindications to interferon and/or ribavirin or their excipients
* Known abuse of alcohol, drugs or pharmaceuticals.
* History, signs or symptoms of a cardiac disease.
* Presence of an implantable pacemaker.
* Any metal implants within the treatment areas (close to the right and/or left deltoid muscles).
* Diagnoses of a serious psychiatric illness which may influence study participation.
* Female subject who is pregnant or breast feeding.
* Female subject not clinically sterile (hysterectomy, tubal ligation or postmenopausal (amenorrhea > 1 year and FSH > 30 mU/ml) OR if not clinically sterile unwilling to use a reliable contraception method.
* Female subject with a positive urine pregnancy test.
* Male subject unwilling to use condom for active prevention of pregnancy from first vaccination to 4 months after last injection.
* Subject or their immediate families being an investigator or site personnel directly affiliated with this study. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Early viral kinetics - Second phase slope of viral decline | 0-4 weeks after SOC onset
Rapid Viral Response (RVR). Percent subjects reaching non-detectable level of HCV-RNA. | 4 weeks after SOC onset
Partial Early Viral Response (pEVR). Percent HCV-RNA positive subjects with more than 2 log 10 decline in HCV-RNA. | 12 weeks after SOC onset
Complete Early Viral Response (cEVR). Percent subjects reaching non-detectable level of HCV-RNA. | 12 weeks after SOC onset

SECONDARY OUTCOMES:
Local tolerance | up to 12 weeks after SOC onset
  Local tolerance will be measured for subjects randomized to vaccination. Local tolerance will be measured 3 times during a time period of 2 h post vaccination. The site of injection will also be inspected at the following visits.
Change from baseline in vital signs | 0 - 12 weeks
Number of patients with AEs | 12 weeks
Change of blood status from baseline | 0 - 12 weeks
Exploratory Analysis - Characterization and quantification of the vaccine primed NS3-immune response | 0 - 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ola RH Weiland, Professor, Principal Investigator — I73 Department of Infectious Diseases, Karolinska Institute, Karolinska University Hospital, Huddinge, Sweden; Anders G Vahlne, Professor, Study Chair — ChronTech Pharma AB, Hälsovägen 7, SE-141 57 Huddinge, Sweden; Matti Sällberg, Professor, Study Director — ChronTech Pharma AB, Hälsovägen 7, SE-141 57 Huddinge, Sweden
Locations (2):
- Sweden (2):
  - I73 Department of Infectious Diseases, Karolinska Institute, Karolinska University Hospital, Huddinge
  - Division of Infectious Diseases, Department of Clinical and experimental medicine, Faculty of Health Sciences, Linköping University, Department of Infectious Diseases, County Council of Östergötland, Linköping